CLINICAL TRIAL: NCT01350050
Title: Topical Pharyngeal Anaesthesia With Articaine for Gastroscopy. A Randomized Double-blind Study on Volunteers
Brief Title: Topical Pharyngeal Anesthesia With Articaine for Gastroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maxim Mazanikov, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: a003c; 2009-011618-12 (EudraCT Number)
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Gastroscopy
Keywords: topical pharyngeal anesthesia; articaine
MeSH Terms: interventions — Carticaine; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- articaine (Active Comparator): Pharyngeal anesthesia with articaine 4% or placebo should randomly and double-blindly applied in turns for every volunteer. In details: 3 ml of Articaine 4%solution or placebo (NaCl 0,9%) will be sprayed into the pharynx 5 minutes before beginning of gastroscopy. Also gastroscope will be lubricated with articaine (or placebo) gel(prepared by adding 4% articaine or 0,9%NaCl in placebo grope to Endopurin® endoscopic lubricant at the day of study).
  Interventions: Drug: articaine
- placebo (Placebo Comparator): Pharyngeal anesthesia with placebo or articaine 4% should be randomly and double-blindly applied in turns for every volunteer. In details: 3 ml of placebo or Articaine 4% solution should be sprayed into the pharynx 5 minutes before beginning of gastroscopy. Also gastroscope will be lubricated with placebo(or articaine) gel(prepared by adding 4% articaine or 0,9%NaCl in placebo grope to Endopurin® endoscopic lubricant at the day of study).
  Interventions: Other: 9% Sodium Chloride solution for injection

INTERVENTIONS:
Drug: articaine — Articaine is intermediate-acting local anesthetic (amide type). Like other local anesthetic drugs, articaine causes a transient and completely reversible state of anesthesia (loss of sensation) during (dental) procedures.
  In dentistry, articaine is used both for infiltration and block injections.
  Other Names: Septocaine; Articadent
  Arms: articaine
Other: 9% Sodium Chloride solution for injection — 9% Sodium Chloride Injection, USP is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection. Each mL contains sodium chloride 9 mg. It contains no bacteriostat, antimicrobial agent or added buffer.
  Other Names: NaCl 0.9%
  Arms: placebo

SUMMARY:
Topical Pharyngeal anesthesia (TPA) is widely used during upper endoscopy. Articaine is local anaesthetic that have not been previously evaluated in pharyngeal anesthesia for upper endoscopy. The aim of this study was to compare pharyngeal anesthesia with 4% articaine to placebo (Na0,9%) during gastroscopy in terms of benefit on patients' and endoscopists' satisfaction.

DETAILED DESCRIPTION:
Topical Pharyngeal anesthesia (TPA) is widely used as an adjunct to sedation during upper endoscopy. TPA improves patient tolerance and the ease of endoscopy.1 Methemoglobinemia and anaphylactic reactions are serious complications of such topical anaesthetic agents, as lidocaine, tetracaine, and benzocaine. Articaine is as a unique amide local anaesthetic that possesses both an amide and an ester linkage and this is of clinical significance in minimizing the risk of overdose (toxic reaction). In routine dental procedures, articaine is a superior anaesthetic to lidocaine. Also, in comparison to lidocaine articaine acts faster and its duration of action is shorter what may be an advantage in such relatively fast procedures as gastroscopy. Articaine have not been previously evaluated in pharyngeal anesthesia for upper endoscopy. The aim of this randomised double-blind placebo controlled study was to compare pharyngeal anesthesia with 4% articaine to placebo (Na0,9%) during gastroscopy in terms of benefit on patients' and endoscopists'satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pregnancy
* allergy to articaine, propofol, alfentanil

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
satisfaction with gastroscopy | one day
  Volunteers were asked to evaluate unpleasantness of gastroscopy (0- most unpleasant, 10-most pleasant), overall satisfaction with gastroscopy (0-extremely dissatisfied 7-extremely satisfied)

SECONDARY OUTCOMES:
vital signs | one day
  Vital signs (heart rate, electrocardiogram, non-invasive blood pressure, peripheral oxygen saturation, end-expiratory carbon dioxide) will be monitored during the gastroscopy and until the discharge.
easiness of gastroscopy performance | one day
  The easiness of gastroscopy performance will be evaluated by endoscopists' with structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Mazanikov, MD, Principal Investigator — Helsinki University Central Hospital,Department of Anesthesiology and Intensive Care; Reino pöyhiä, MD,PhD, Study Director — Helsinki University Central Hospital,Department of Anesthesiology and Intensive Care; Marianne Udd, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Gastrointestinal and General Surgery; Jorma Halttunen, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Gastrointestinal and General Surgery; Leena Kylänpää, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Gastrointestinal and General Surgery; Outi Lindström, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Gastrointestinal and General Surgery; Martti Färkkilä, MD,Professor, Principal Investigator — Helsinki University Central Hospital,Department of Medicine, Division of Gastroenterology
Locations (1):
- Helsiki University Central Hospital,Meilahti Hospital,Endoscopy unit, Helsinki, Uusimaa, Finland